CLINICAL TRIAL: NCT05536310
Title: Trilogy Heart Valve System for Management of Patients With Aortic Valve Disease: Patient Registry and Post-Market Clinical Follow-up Study
Brief Title: TAVIS Registry - Trilogy Heart Valve System for Management of Patients With Aortic Valve Disease
Acronym: TAVIS
Status: Not yet recruiting | Type: Observational
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-0099
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Regurgitation; Aortic Valve Stenosis With Insufficiency; Constriction, Pathologic; Aortic Valve Disease; Heart Valve Diseases; Cardiovascular Diseases in Old Age; Ventricular Outflow Obstruction; Aortic Stenosis, Severe
Keywords: Trilogy; Aortic Valve Disease; Transcatheter aortic valve replacement (TAVR); Aortic Valve Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Constriction, Pathologic; Aortic Valve Disease; Heart Valve Diseases; Ventricular Outflow Obstruction | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Trilogy TAVI: Patients receiving JenaValve Trilogy Heart Valve System for management of symptomatic, severe aortic stenosis (AS)/ aortic regurgitation (AR) who are at high risk for surgical aortic valve replacement (SAVR)
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — TAVI with the JenaValve Trilogy Heart Valve System

SUMMARY:
To collect information about the management of symptomatic severe Aortic Stenosis (AS) and Aortic Regurgitation (AR) using transcatheter aortic valve replacement (TAVI).

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a narrowing of the aortic valve opening causing restricted blood flow from the left ventricle to the aorta and may also affect the pressure in the left atrium. Aortic regurgitation (AR) is a condition where the aortic valve in the heart does not close tightly and allows some blood to leak back into the heart chamber. Symptoms of AS and AR may include fatigue and shortness of breath. Aortic valve disease can affect both elderly and younger populations. TAVIS Registry will collect data from patients suffering from either AS or AR using a minimally invasive transcatheter aortic valve implantation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed ICF and are indicated by their doctors to be treated with Trilogy Heart Valve System in line with the medical standard of care
2. Patients with symptomatic severe aortic regurgitation (AR) or symptomatic, severe aortic stenosis (AS), who are at high risk for SAVR as documented by the heart team and Heart Team agrees that patient can undergo SAVR for "bail out"/to address unfavorable circumstances if necessary
3. Patients 18 years of age or older
4. Patient is willing to participate in the study, provides signed Informed Consent/Data Authorization Form and authorizes the sharing of data in the study
5. The subject and treating physician agree the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Patients who have known hypersensitivity or contraindication to Nitinol (titanium and/or nickel), an anti-coagulation/anti-platelet regimen or contrast medium that cannot be managed with premedication
2. Patients who have active bacterial endocarditis or other active infections
3. Pediatric (<18 years) and/or pregnant/nursing patients
4. Congenital/functional unicuspid, bicuspid or quadricuspid native aortic valve morphology
5. Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
6. Echocardiographic evidence of current left heart thrombus
7. Hypertrophic cardiomyopathy with or without obstruction.
8. Access vessel characteristics that would preclude safe placement of the JenaValve 20Fr introducer sheath, such as severe obstructive calcification, severe tortuosity, or vessel diameter <7mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic severe aortic regurgitation or symptomatic severe aortic stenosis undergoing treatment with JenaValve Trilogy Heart Valve System
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30-days post-index procedure
  Mortality from any cause in patients receiving TAVI for AR or AS

SECONDARY OUTCOMES:
Death | 1 year
  Reported death in patients participating in TAVIS Registry
Stroke | 30 days and 1 year
  Reported stroke in patients participating in TAVIS Registry
Major vascular complications | 30 days
  Reported vascular complications in patients participating in TAVIS Registry
Major and life-threatening bleeding | 30 days
  Reported major and life-threatening bleeding complications in patients participating in TAVIS Registry
New conduction defects requiring permanent pacemaker | 30 days
  Reported conduction defects requiring permanent pacemaker in patients participating in TAVIS Registry
Acute kidney injury stage 2-3 | 7 days
  Reported kidney injury complications in patients participating in TAVIS Registry
New onset atrial fibrillation | 30 days
  Reported new onset atrial fibrillation in patients participating in TAVIS Registry

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Baldus, MD, Principal Investigator — University Hospital of Cologne Heart Center; Hendrik Treede, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (3):
- Germany (3):
  - Herz-und Diabeteszentrum NRW Ruhr-Universität Bochum Bad Oeynhausen, Bad Oeynhausen
  - University Hospital of Cologne Heart Center, Cologne
  - University Hospital Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoghbi WA, Adams D, Bonow RO, Enriquez-Sarano M, Foster E, Grayburn PA, Hahn RT, Han Y, Hung J, Lang RM, Little SH, Shah DJ, Shernan S, Thavendiranathan P, Thomas JD, Weissman NJ. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2017 Apr;30(4):303-371. doi: 10.1016/j.echo.2017.01.007. Epub 2017 Mar 14. No abstract available. PMID 28314623
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Jun 20;135(25):e1159-e1195. doi: 10.1161/CIR.0000000000000503. Epub 2017 Mar 15. No abstract available. PMID 28298458
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Hamid N, Ranard LS, Khalique OK, Hahn RT, Nazif TM, George I, Ng V, Leon MB, Kodali SK, Vahl TP. Commissural Alignment After Transfemoral Transcatheter Aortic Valve Replacement With the JenaValve Trilogy System. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2079-2081. doi: 10.1016/j.jcin.2021.07.025. No abstract available. PMID 34556282
- [Background] Treede H, Rastan A, Ferrari M, Ensminger S, Figulla HR, Mohr FW. JenaValve. EuroIntervention. 2012 Sep;8 Suppl Q:Q88-93. doi: 10.4244/EIJV8SQA16. PMID 22995119
- [Background] Poschner T, Werner P, Kocher A, Laufer G, Musumeci F, Andreas M, Russo M. The JenaValve pericardial transcatheter aortic valve replacement system to treat aortic valve disease. Future Cardiol. 2022 Feb;18(2):101-113. doi: 10.2217/fca-2021-0065. Epub 2021 Oct 14. PMID 34647465
- [Background] Ng VG, Khalique OK, Nazif T, Patel A, Hamid N, George I, Bapat V, Hahn R, Kodali S, Vahl TP. Treatment of Acute Aortic Insufficiency With a Dedicated Device. JACC Case Rep. 2021 Mar 24;3(4):645-649. doi: 10.1016/j.jaccas.2021.01.021. eCollection 2021 Apr. PMID 34317595